CLINICAL TRIAL: NCT06193902
Title: A Phase I/IIa Open-label Dose Escalation Trial Evaluating the Safety and Preliminary Efficacy of LEU011 in Subjects With Relapsed/Refractory Solid Tumours
Brief Title: LEU01101: Safety and Preliminary Efficacy of LEU011 in Solid Tumours.
Acronym: AERIAL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leucid Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LEU01101
Record Dates: First submitted 2023-12-12; First posted 2024-01-05 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Tumor, Solid
Keywords: Solid Tumours, NKG2D Ligands, Adult
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LEU011 (Experimental): Infusion of target dose of LEU011
  Interventions: Biological: LEU011

INTERVENTIONS:
Biological: LEU011 — Immunotherapy

SUMMARY:
This is a dose-escalation open-label Phase 1/2a study. The purpose of this first-in-human study is to assess the safety and tolerability of LEU011 (autologous CAR T cells targeting NKG2D ligands) in patients with solid tumours.

DETAILED DESCRIPTION:
This is a dose-finding study of the investigational immunotherapy LEU011 in patients with NKG2DL-expressing solid tumours. The study will assess the safety and tolerability of LEU011 and is designed to determine the maximum tolerated dose (MTD) of LEU011.

Enrolled patients will undergo a whole blood procurement in order to manufacture LEU011. Subjects will receive LEU011 as a single IV dose following pre-conditioning chemotherapy and will be followed up for up to two years on this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed solid tumour.
2. 18 years or older at time of consent
3. Relapsed/refractory solid tumour with no standard treatment options available or suitable (e.g. hypersensitivity reaction) and no curative approach possible.
4. Tumour expression of NKG2DL protein. The minimum requirement is the presence of one or more ligands on 10% or more cells, encompassing tumour and/ or stroma.
5. At least one target lesion measurable by RECIST v1.1 criteria on CT or MRI scanning
6. Eastern Co-operative Oncology Performance Status of 0-1.
7. Normal cardiac function as assessed by electrocardiography and echocardiography (ECHO. Left ventricular ejection fraction must be normal according to institutional values.
8. Baseline oxygen saturation of at least 95%
9. Haematology results must show:

   * neutrophils >1.5 x 109/L,
   * platelets >100 x 109/L,
   * haemoglobin >90g/L,
   * INR <1.3.
   * Lymphocytes >0.4 x 109/L
10. Biochemistry results must show:

    * creatinine clearance > 40 mL/min/1.73 m2 (calculated using the Chronic Kidney Disease Epidemiology [CKD-EPI] equation); bilirubin <1.25 times ULN;
    * ALT/ AST <2.5 times ULN (<5 times ULN if liver metastases present);
    * Albumin > 30g/L
11. Agree to use highly effective contraception (if applicable). Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test.
12. Disease amenable to biopsy.
13. Life expectancy of at least 6 months, in the investigator's opinion.
14. Written informed consent prior to any trial procedure and registration.
15. Subjects must agree to participate in an additional LTFU trial for up to 15 years after completion of this trial.

Exclusion Criteria:

1. Subjects with HIV-1, HIV-2, HTLV-1, HTLV-2, active Hepatitis B, active Hepatitis C, or active Syphilis infection. Subjects without active Hepatitis B infection who are anti-core antibody positive can be considered for recruitment subject to suitability to receive nucleoside or nucleotide analogue prophylaxis.
2. Subject must not have received any anti-cancer treatment within 28 days of lymphodepletion (prior to LEU011). This criterion applies to the following additional therapies: (i) systemic corticosteroids (> 20mg prednisolone/ day); (ii) any other systemic immunomodulatory agent (but see 11 below); (iii) radiotherapy; (iv) chemotherapy; (v) endocrine therapy or (vi) any investigational medicinal product.
3. Regarding (iv) Chemotherapy: Interval is extended to 6 weeks in the case of nitrosoureas. This criterion does not apply to the use of lymphodepleting chemotherapy prior to treatment with LEU011.
4. Prior LEU011 therapy. However, prior immune checkpoint blockade (e.g. anti-PD1, PD-L1 or CTLA-4) or immune agonist antibody therapy (e.g. anti-4-1BB, OX40, CD40 etc) does not preclude participation, but there must be a washout period of 30 days prior to treatment with LEU011.
5. Concurrent use of warfarin anticoagulant therapy and other coumarins is not permissible. Other classes of anticoagulant can be given.
6. The presence of major co-morbidity such as active major medical illness of the cardiovascular, respiratory or immune system that is likely to impair ability to undergo trial therapy, such as recent myocardial infarction, congestive cardiac failure, active gastrointestinal bleeding, active gastrointestinal ulceration, inflammatory bowel disease, ischaemic heart disease, peripheral arterial disease, pneumonitis, intestinal obstruction, sepsis or uncontrolled hypertension.
7. Clinically active autoimmune disease e.g., coeliac disease (an abnormal TTG antibody test precludes recruitment) or interstitial lung disease. Sub-clinical or quiescent autoimmune disease does not exclude from participation (e.g. euthyroid patients on thyroxine replacement therapy or patients with type 1 diabetes on insulin therapy).
8. Active infection that requires antimicrobial treatment.
9. Subjects who, in the Investigator's judgement, are unlikely to complete or comply with all protocol required study visits or procedures.
10. Hypersensitivity to any component of LEU011 (e.g. Albumin or DMSO allergy).
11. Cyclophosphamide or fludarabine allergy or contraindication.
12. Pregnancy.
13. Breastfeeding.
14. Subjects who have received a live vaccine four weeks or fewer before enrolment are ineligible for recruitment to the study. During treatment and for three months after treatment with fludarabine, administration of live vaccines is prohibited. None of the currently available covid 19 vaccines are considered to be live for this purpose since all are replication defective.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate the dose limiting toxicity, safety and tolerability of a single dose of LEU011 in subjects with NKG2DL expressing relapsed/refractory solid tumours | 28 days post administration of LEU011 immunotherapy
  Incidence and nature of dose limiting toxicities will be graded by American Society of Transplantation and Cellular Therapy (ASTCT) consensus criteria.
To identify a recommended Phase 2 dose (RP2D) of LEU011 | 28 days post administration of LEU011 immunotherapy
  RP2D will be the MTD.

CONTACTS AND LOCATIONS:
Overall Officials: John Maher, Study Chair — Leucid Bio
Locations (2):
- United Kingdom (2):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No